CLINICAL TRIAL: NCT07131267
Title: Evaluating Sexual Functioning in Trans Men During the Gender Affirmation Process: A Mixed Methods Study
Acronym: ESFTMGAP
Status: Recruiting | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Imran Gokcen Yilmaz-Karaman, Associate professor doctor, Eskisehir Osmangazi University
Other Study IDs: EskisehirOU 28.05.2025/26
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Sexual Functioning; Transgender Men; Gender Affirmation Surgery
Keywords: sexual functioning; transgender men; gender affirmation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Trans men during the gender affirmation process

SUMMARY:
Both sexual experiences and the process of gender transition initiated to reduce gender dysphoria carry cultural characteristics. Gender categories, societal expectations for each gender, and attitudes toward sexual minorities in a given society can shape the lived experiences of trans individuals. Therefore, research on individuals with gender dysphoria in different cultural contexts is of great importance. To our knowledge, no study in Türkiye has examined sexual functioning in trans individuals undergoing gender transition. For this reason, our study aimed to investigate how sexual functioning is affected by the gender transition process in trans men with gender dysphoria, using both quantitative and qualitative methods.

DETAILED DESCRIPTION:
For the quantitative part of the study, 52 participants will receive a sociodemographic and clinical data form, Arizona Sexual Experiences Scale, Sexual Desire Inventory, Utrecht Gender Dysphoria Scale, Depression Anxiety Stress Scale-21, and WHOQOL-100 sexual quality of life subscale.

While performing a qualitative study, 12 participants will receive questions about their sexual functioning during the gender affirmation process.

ELIGIBILITY:
Inclusion Criteria:

18 years or older Diagnosed with gender dysphoria by two different physicians Getting medical support for the gender affirmation process

Exclusion Criteria:

Over 65 years Diagnosed with intellectual disability, dementia, or organic mental disorders Having a systemic disease that negatively impacts sexual function Getting a score above 3 on the Clinical Global Impression Scale

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans men during the gender affirmation process
Study Population: Trans men during the gender affirmation process
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sexual functioning | Day 1
  Arizona Sexual Experience Scale: It is designed to measure five specific items identified as fundamental elements of sexual function. The scale was designed by McGahuey (McGahuey et al., 1997). The Turkish validity and reliability of the scale was conducted by Atilla Soykan (Soykan, 2004). Higher scores indicate higher levels of dysfunction.
Sexual desire | Day 1
  Sexual Desire Inventory-2: It is a 14-item, self-administered questionnaire measuring sexual desire (Spector et al., 1996). It includes subscales of sexual motivation, sexual satisfaction, sexual relationship quality, activity frequency, and behavioral diversity to capture the multidimensional nature of sexual desire. The Turkish validity and reliability of the scale, along with other languages, were conducted in Castro-Calvo's study (Castro-Calvo et al., 2024). High scores indicate high sexual desire.

CONTACTS AND LOCATIONS:
Overall Officials: Imran G Yilmaz-Karaman, Assoc.Prof., Study Director — Eskişehir Osmangazi University, Faculty of Medicine
Locations (1):
- Eskişehir Osmangazi University, Faculty of Medicine, Department of Psychiatry, Eskişehir, Türkiye, Turkey (Türkiye)